CLINICAL TRIAL: NCT00311493
Title: A Phase IV, Randomized, Open-Label, Multi-Center Study in Adults: Evaluation of Long-Term Immunogenicity in Subjects Boosted With a New TBE Vaccine for Adults (Free of Protein-Derived Stabilizer) in Study V48P2E1, 5 Years After First Booster Immunization and Evaluation of Booster Kinetics in Subjects Boosted With a New TBE Vaccine for Adults (Free of Protein-Derived Stabilizer), 5 Years After First Booster Immunization
Brief Title: Evaluation of Long-Term Immunogenicity in Subjects Boosted With a TBE Vaccine for Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: V48P2E3; 498
Record Dates: First submitted 2006-04-03; First posted 2006-04-06 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Encephalitis, Tick-Borne
Keywords: TBE; vaccine; adults
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: Tick-Borne Encephalitis vaccine

SUMMARY:
The purpose of this study it is to evalutate the persistence of antibodies after a booster immunisation with a TBE vaccine for adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged >18 who participated in another study on TBE vaccination

Exclusion Criteria:

* Subjects with any condition, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179
Dates: Start 2006-02

PRIMARY OUTCOMES:
Long-term antibody kinetics as measured both by ELISA and neutralisation test (NT) five years after first booster immunization.

SECONDARY OUTCOMES:
Booster response in a subset of subjects as measured by NT, ELISA and cellular immunity on Days 3, 5, 7 and 21 after 2nd booster immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Drug Information Services, Study Director — Chiron Corporation
Locations (1):
- Regensburg, Germany